CLINICAL TRIAL: NCT07161050
Title: Effects of a Low Nicotine Standard and Tobacco Prices on Illegal Cigarette Purchasing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VT IRB #25-813; 5P01CA200512 (NIH)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking; E-cigarette Use
Keywords: Experimental Tobacco Marketplace; Illegal cigarette
MeSH Terms: conditions — Cigarette Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: Participants will complete one ETM session with a total of 18 purchasing trials, 9 trials in each of the two conditions - NNC and VLNC. The participant's preferred cigarette will be available in both the LETM and iETM in the NNC condition. In the VLNC condition, the preferred cigarette will be available only in the iETM and VLN cigarettes will be available in the LETM. E-cigarettes, nicotine replacement therapy, snus, and nicotine pouches will be available throughout all trials in the LETM. Within each condition, we will manipulate the price of illegal cigarettes (1xMP, 1.5x MP, 2x MP). At each level of illegal cigarette price, we will also manipulate the price of NVP (1/2x MP, 1x MP, 2x MP). This design will permit the investigation and comparison of the effects of a VLNC standard as well as changes in illegal and NVP price. The investigators will counterbalance the order of the conditions within the ETM session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive cigarette smokers (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to all of the conditions described in the intervention section.
  Interventions: Behavioral: Nicotine Content; Behavioral: Illegal cigarette price; Behavioral: E-cigarette price
- Dual cigarette/ nicotine vaping product users (Experimental): Dual cigarette and nicotine vaping product users will be recruited and will be exposed to all of the conditions described in the intervention section
  Interventions: Behavioral: Nicotine Content; Behavioral: Illegal cigarette price; Behavioral: E-cigarette price

INTERVENTIONS:
Behavioral: Nicotine Content — In the full nicotine conditions, participants' preferred cigarettes and NVP products will be available in the LETM and preferred cigarettes will be available in the iETM. In the low nicotine conditions, a ban will permit only VLNCs in the LETM and preferred cigarettes will be available in the iETM.
  Other Names: very-low nicotine standard
Behavioral: Illegal cigarette price — At each level of nicotine content, we will manipulate the price of illegal cigarettes (1xMP, 1.5x MP, 2x MP). MP is market price.
Behavioral: E-cigarette price — At each level of nicotine content and illegal cigarette price, we will manipulate the price of e-cigarettes (1xMP, 1.5x MP, 2x MP). MP is the market price.

SUMMARY:
This study will investigate the effects of a very-low-nicotine cigarette (VLNC) standard, e-cigarette price, and illegal cigarette price on illegal product purchasing and alternative product use in a virtual marketplace.

DETAILED DESCRIPTION:
This experiment will examine the effects of a VLNC standard, electronic cigarette price, and illegal cigarette price on illegal cigarette purchasing. Exclusive cigarette smokers and dual cigarette/nicotine vaping product (NVP) users, stratified by age, will complete multiple scenarios in the legal Experimental Tobacco Marketplace. The investigators will examine the effects of a VLNC standard, predicted to promote illegal purchasing. In the NNC conditions, participants' preferred normal nicotine content (NNC) cigarettes, NVPs, and a variety of other products will be available in the ETM, and preferred NNC cigarettes will also be available in the illegal marketplace. In the VLNC standard conditions, a ban will permit only VLNCs legally in the ETM, but preferred NNC cigarettes will continue to be available illegal marketplace. In this experiment, which will be completed in the lab, we will test three levels of NVP prices and three levels of illegal cigarette prices in scenarios under a VLNC standard or NNC condition. This study will involve a total of three sessions, including an assessment session, an ETM session, and a follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent Be at least 21 years of age or older Provide a breath sample for measuring carbon monoxide (CO ≥ 8 ppm) Stable tobacco use patterns for at least two months

Exclusion Criteria:

For exclusive cigarette smokers:

Smoke at least 10 cigarettes daily and do not use NVPs regularly (no more than 9 times in the last month).

For dual cigarette/NVP users:

Smoke at least 10 cigarettes daily and use NVPs at least 3 times in a week (report use of closed nicotine salt system)

For both groups:

Have plans to move out of the area Have a serious or unstable physical or mental health condition Taking a tobacco cessation medication or medication that interferes with nicotine metabolism, motivation or reinforcement Report concrete, immediate plans to alter/quit using their usual nicotine products at the beginning of the study Being pregnant or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Percent of budget allocated to each product category (eg, legal cigarettes, e-cigarettes, illegal cigarettes, etc) in the marketplace | 1 day
  The investigators will measure the percent of each partcipants' study budget spent on products from each category (eg, legal cigarettes, e-cigarettes, illegal cigarettes, etc) in the marketplace

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Freitas-Lemos, PhD, Principal Investigator — Fralin Biomedical Research Institute at Virginia Tech Carilion
Locations (1):
- Fralin Biomedical Research Institute at Virginia Tech Carilion, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.